CLINICAL TRIAL: NCT05193474
Title: Evaluate Serious Illness Treatment Preferences and Outcomes in the Patients Receiving Peritoneal Dialysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 202106064RINB
Record Dates: First submitted 2021-12-08; First posted 2022-01-18 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2021-08

CONDITIONS: ESRD; Peritoneal Dialysis
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Refuse to integrate palliative care into usual care. (No Intervention): Usual ESRD care team
- Agree to integrate palliative care into usual care. (Experimental): Usual ESRD care + combined palliative care team
  Interventions: Behavioral: integrated palliative care

INTERVENTIONS:
Behavioral: integrated palliative care — shared decision making with patient, and timely integrated palliative care according to patient's preference
  Arms: Agree to integrate palliative care into usual care.

SUMMARY:
The goal of this clinical research study is to study the cardiopulmonary resuscitation (CPR) preferences of patients receiving peritoneal dialysis and how these preferences are associated with their responses to questions about aspects of end-of-life care.

This prospective cohort clinical trial aims to provide evidence on the preferences of end of life care in patients receiving peritoneal dialysis, thereby provide optimal care according to patients' preferences and choices through effective communication and clear goals of care.

DETAILED DESCRIPTION:
This is a prospective cohort study to survey cardiopulmonary resuscitation (CPR) preferences of patients receiving peritoneal dialysis and how these preferences are associated with their responses to questions about aspects of end-of-life care for end stage renal disease(ESRD) patients, and actively survey their palliative care need to share decision making with ESRD patient whether to receive standardized palliative care interventions by the interdisciplinary palliative care team, including treatment of suffering symptoms, non-pharmacologic therapies. The investigators will enroll 500 patients. The eligibility criteria are shown later part. After obtaining consent from the patient, the investigators will conduct baseline assessments and start the patient on a 10minutes questionnaire. The questionnaire was cited from 2016-CA-POLST, which is in Chinese version for better understanding. POLST is an approach to end-of-life planning based on conversations between patients, loved ones, and health care professionals designed to ensure the patient only receive the care that patients themselves wish to. After that, the investigators will active survey the patient who had higher mortality rate within one year by using 1. Palliative Care Screening Tool (PCST)， 2."Surprise" Question，3. Integrated model risk≥10%. For the patient who had higher mortality rate within one year (>10%), the investigators would evaluate the degree of symptoms burden by using ESAS-r: Renal. For the patient who had moderate to severe symptoms burden, the investigators would share decision making with them to discuss whether to receive combined palliative care. The investigators would divide the patients to two group according to patient decision. (1) Usual ESRD care team (2) Usual ESRD care + combined palliative care team. And the investigators would compare the quality of life and quality of death, and symptoms burden after 3/6/12 months receiving timely integrated palliative care to the other group Evaluate outcomes including quality of life (EQ-5D-5L), quality of death (GDS), symptoms burden(ESAS-r:Renal)

ELIGIBILITY:
Inclusion Criteria:

1. [Patients] Diagnosis of ESRD
2. [Patients] Under treatment of peritoneal dialysis
3. [Patients] Age 20 years or older
4. [Caregivers] Age20 years or older

Exclusion Criteria:

* [Patients] unable to understand or fill in the questionnaire

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-02-01 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
the preferences of end of life care in patients receiving peritoneal dialysis | up to 24 weeks
  Participants were asked to respond to the questions(POLST questionnaire) associated to life-sustaining treatment preference including CPR preference and other treatment preferences, and life values,

SECONDARY OUTCOMES:
compare the quality of life after receiving timely integrated palliative care to the other group | 3 moths,6 months and 12months after receiving timely integrated palliative care
  Quality of life(The EuroQol-5 Dimension 5-level (EQ-5D-5L)) The EQ-5D instrument is the most widely used generic preference-based measure of health.
  The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
compare the quality of death after receiving timely integrated palliative care to the other group | 3 moths,6 months and 12months after receiving timely integrated palliative care
  Quality of death(Good Death Scale (GDS)) Good Death Scale (GDS) is a provider assessment scale of the quality of dying of terminally ill patients. It contains 5 items including the awareness that one is dying (0 = complete ignorance, 3 = complete awareness), accepting death peacefully (0 = complete unacceptance, 3 = complete acceptance), propriety (0 = no reference to the patient's will, 1 = following the family's will alone, 2 = following the patient's will alone, 3 = following the will of both the patient and their family), death timing (0 = no preparation, 1 = the family alone had prepared, 2 = the patient alone had prepared, 3 = both the patient and their family had prepared), and degree of physical comfort (0 = a lot of suffering, 1 = suffering, 2 = a little suffering, 3 = no suffering). The score ranges from 0 to 15.
compare the symptoms burden after receiving timely integrated palliative care to the other group | 3 moths,6 months and 12months after receiving timely integrated palliative care
  Symptoms burden(Edmonton Symptom Assessment System. Revised Renal (ESAS-r:Renal)) The ESAS-r helps to assess nine common symptoms in palliative care patients. The ESAS-r is one valuable part of a holistic clinical assessment. It is not a complete assessment in itself. The patient should be instructed to rate the severity of each symptom on a 0 to 10 scale, where 0 represents absence (or best possible intensity) of the symptom and 10 represents the worst possible severity. The number should be circled on the scale.
  The circled numbers can be transcribed onto the ESAS-r graph. The patient should be instructed to rate each symptom according to how s/he feels now. The health care professional may choose to ask additional questions about the severity of symptoms at other time points (e.g. symptom severity at best and at worst over the past 24 hours)
compare the ICU admission frequency after receiving timely integrated palliative care to the other group | 3 moths,6 months and 12months after receiving timely integrated palliative care
  ICU admission frequency

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Fu Lai, M.d., Principal Investigator — National Taiwan University Hospital